CLINICAL TRIAL: NCT07047625
Title: The Application Effect of Health Education Path Nursing Program in Patients After Percutaneous Nephrolithotomy
Brief Title: The Application of Health Education Path Nursing Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuyang Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Antao Dong, Resident Physician, Fuyang Affiliated Hospital of Anhui Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FuyangH002
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Nephrolithiasis
Keywords: Nephrolithiasis; Percutaneous nephrolithotripsy; Health education path
MeSH Terms: conditions — Nephrolithiasis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Behavioral: control group (Routine nursing)
- experimental group (Experimental)
  Interventions: Behavioral: Experimental group （Health education path）

INTERVENTIONS:
Behavioral: control group (Routine nursing) — the implementation of routine treatment and nursing measures, including (1) Monitoring vital signs: according to the condition of vital signs change detection, found abnormal, timely notify the doctor, comply with medical treatment, observe the curative effect. (2) Relieve pain: tell patients the method of distraction, follow the doctor's advice, and observe the curative effect. (3) Improve disease awareness: Inform patients or family members of disease-related knowledge, examination, diagnosis and treatment, surgery and other purposes, significance and precautions. (4) Ensure patient safety: strengthen safety education, strict three check seven pairs, bed placed a variety of safety warning signs. (5) Avoid the occurrence of unexpected risks: guide patients and their families to prevent burns, trauma, etc. (6) Prevention of infection: strict implementation of disinfection and isolation system, the implementation of hand hygiene norms, reduce visits. (7) Raise the affected limb, early f
  Arms: control group
Behavioral: Experimental group （Health education path） — On the basis of the control group, the health education path nursing program was adopted. The specific intervention measures were as follows: ① A program implementation team was set up, including 2 urologists, 2 nurses and 1 psychological counselor. All members have received relevant professional training; ②Two nurses were the main liaisons for the intervention and were responsible for monitoring the treatment and nursing of patients throughout the course. The workflow was as follows: starting from the patient's discomfort experience, the patient was managed according to the nursing procedure steps. By assessing the patient's existing discomfort symptoms, interventional cognitive intervention and psychological intervention, and based on the intervention plan proposed in this study, a health education path nursing plan was developed for patients from the aspects of diet, liquid intake, position adjustment, and symptomatic intervention (see Table 1). In the process of intervention, feedb
  Arms: experimental group

SUMMARY:
Objective: To explore the effect of health education pathway on self-management ability and quality of life of patients after percutaneous nephrolithotomy. Method: Patients who underwent renal calculi in our hospital from January 1,2023 to August 31,2023 were collected by convenient sampling method. According to the order of enrollment, they were divided into control group and experimental group. Self-management indicators and quality of life indicators were collected for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients with preoperative urinary tract infection received anti-infective treatment and were well controlled;
* The levels of blood pressure, blood glucose and electrolyte abnormalities found before operation returned to normal and remained stable after active treatment by doctors;
* Patients undergoing percutaneous nephrolithotripsy.

Exclusion Criteria:

* There were systemic hemorrhagic diseases, and the coagulation function has not been corrected;
* Long-term use of anticoagulant drugs such as aspirin, warfarin, preoperative non withdrawal for more than 1 week;
* Renal malignant tumor, pelvic ectopic kidney, polycystic kidney and severe renal prolapse were found before operation;
* Pregnancy patients;
* Uncontrolled urinary tract infection;
* Infectious disease activity period, such as tuberculosis, hepatitis and other patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
The self-management ability of the two groups of subjects | three months
  The self-management ability refers to the ' self-management ability survey scale for patients with urinary calculi ' in the study of Wang Hongdan et al. The Likert5 score method was used to evaluate the self-management ability of the two groups of patients before and three months after the intervention from the five dimensions of diet control, proper exercise, emotional management, medication compliance and regular follow-up. The total score was 5-25 points. The higher the score, the stronger the patient's self-management ability.
The quality of life of the two groups of subjects | Three months
  SF-36 was used as a quality of life questionnaire. It comprehensively summarized the quality of life of respondents from eight aspects: physiological function, physiological function, physical pain, general health status, energy, social function, emotional function and mental health. The higher the score, the better the situation

CONTACTS AND LOCATIONS:
Locations (1):
- the Fuyang Affiliated Hospital of Anhui Medical University, Fuyang, Anhui, China

IPD SHARING:
Plan to Share IPD: No